CLINICAL TRIAL: NCT00556127
Title: Programma di Terapia Per Pazienti Affetti da Linfoma Diffuso a Grandi Cellule B CD20 Positive
Brief Title: Rituximab in Addition to Chemotherapy With Autologous Stem Cell Transplantation as Treatment Diffuse Large B-Cell Lymphoma
Acronym: DLBCL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Italiano Multiregionale per lo studio dei Linfomi e delle Leucemie (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMURELL-DLBCL; Eudract Number 2004-000543-19
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2007-11-09 (Estimated); Status verified 2007-11

CONDITIONS: Diffuse Large B-Cell Lymphoma; POOR PROGNOSIS
Keywords: Large B-cell Lymphoma; Rituximab; ASCT
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Epirubicin; Cyclophosphamide; Vincristine; Prednisone; Granulocyte Colony-Stimulating Factor; Mitoxantrone; Dexamethasone; Carmustine; Etoposide; Melphalan; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Rituximab; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Vincristine; Drug: Prednisone; Drug: Granulocyte-colony-stimulating factor; Drug: Mitoxantrone; Drug: Cytarabine ARA-C; Drug: Dexamethasone; Drug: Carmustine BCNU; Drug: Etoposide; Drug: Melphalan; Radiation: Radiotherapy; Procedure: PBSC reinfusion

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 on day 1
Drug: Epirubicin — 110 mg/m2 on day 3
Drug: Cyclophosphamide — 1200 mg/m2 on day 3
Drug: Vincristine — 1.4 mg/m2 (maximum 2 mg) on day 3
Drug: Prednisone — 40 mg/m2 from day 1 to 5
Drug: Granulocyte-colony-stimulating factor — (G-CSF 5 μg/Kg/day) from day 5 to day 11
Drug: Mitoxantrone — 8 mg/m2 for 3-day
Drug: Cytarabine ARA-C — 2 g/m2/12 hours for six doses in 3-hour infusion
Drug: Dexamethasone — 4 mg/m2/12 hours before ARA-C administration
Drug: Carmustine BCNU — 300 mg/m2 on day -7
Drug: Etoposide — 100 mg/m2/12 hours
Drug: Melphalan — 140 mg/m2 on day -2
Radiation: Radiotherapy — Involved Field Radiotherapy (IF-RT)
Procedure: PBSC reinfusion — ASCT

SUMMARY:
The purpose of this trial was to evaluate efficacy and safety of adding Rituximab to dose-dense and High-Dose Chemotherapy (HDC) with Autologous Stem Cell Transplantation (ASCT) as first line treatment in young patients with DLBCL at Intermediate-High and High risk aaIPI score

ELIGIBILITY:
Inclusion Criteria:

* previously untreated aggressive B-cell lymphoma (Diffuse Large B-Cell,
* Primary Mediastinal,
* Follicular grade III b Lymphoma);
* age 18 to 60;
* III-IV Ann Arbor stage;
* 0-2 Eastern Cooperative Oncology Group (ECOG) performance status (PS);
* intermediate-high (IH) and high (H) risk score according to age-adjusted International Prognostic Index (IPI).
* Patients with Primary Mediastinal Lymphoma were included only if they had advanced stage III or IV disease.

Exclusion Criteria:

* HIV,
* hepatitis B or C virus seropositivity;
* CNS involvement at diagnosis;
* abnormal renal, pulmonary and hepatic function;
* left ventricular ejection fraction less than 45%;
* pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2002-06; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Failure-free survival | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Vitolo, MD, Principal Investigator — S.C. Ematologia II - OSP.S. GIOV.BATTISTA MOLINETTE - TORINO (TO) -
Locations (14):
- Italy (14):
  - Az. Ospedaliera SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Ospedale Regionale, Divisione di Oncologia,, Aosta
  - Azienda Ospedaliera Ospedale Policlinico Consorziale, Bari
  - Osp. degli Infermi, Biella
  - Spedali Civili, Brescia
  - Centro Trapianti Midollo Osseo, P.O. Businco, Cagliari
  - Ospedale S. Gerardo, Monza
  - Osp. maggiore della Carità, Novara
  - Università degli Studi Policlinico Monteluce, Perugia
  - Divisione di Medicina, Ospedale Generale E. Agnelli, Pinerolo, Torino
  - Istituto per la Ricerca e la Cura del Cancro, Candiolo, Torino
  - Osp. S. Giovanni Battista "Molinette", Torino
  - Ospedale di Chivasso e Ivrea, Torino
  - Stabilimento Ospedaliero Ciriè -, Torino